CLINICAL TRIAL: NCT02721641
Title: A Single Arm, Multi-Center, International, Continuation Trial of Recombinant Humanized Antibody Herceptin (Trastuzumab) in Patients With HER2-Overexpressing Tumors
Brief Title: A Continuation Study of Herceptin (Trastuzumab) in Participants With Metastatic or Locally Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO15943; 2007-000348-28 (EudraCT Number)
Record Dates: First submitted 2016-03-24; First posted 2016-03-29 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Trastuzumab

ARMS (1):
- Herceptin (Experimental): Participants with stable disease and HER2-overexpressing metastatic or locally advanced cancer will receive expanded access to IV Herceptin until disease progression, unacceptable toxicity, death, or decision by the investigator or participant to discontinue treatment.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be administered as either 2 milligrams per kilogram (mg/kg) once weekly (first dose as a 4-mg/kg loading dose) or 6 mg/kg every 3 weeks (first dose as an 8-mg/kg loading dose) via IV infusion over 90 minutes.
  Other Names: Trastuzumab

SUMMARY:
This study is designed to provide continued access to intravenous (IV) Herceptin and to evaluate long-term outcomes and overall safety in participants with stable disease and human epidermal growth factor 2 (HER2)-overexpressing metastatic or locally advanced cancer who have completed a prior study with IV Herceptin.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing participants from any completed global Roche-sponsored Herceptin trial
* Participants enrolled in any Roche-sponsored Herceptin trial who have at least stable disease (or whose disease has not recurred) during Herceptin therapy at the end of the lead-in trial
* Available study termination data (including tumor assessment and laboratory data) on the Case Report Form for the lead-in trial
* Judged eligible by the investigator following a thorough risk/benefit assessment, if signs of chronic heart failure developed during the lead-in trial

Exclusion Criteria:

* Pregnant or nursing women
* Women of childbearing potential unless using effective contraception as determined by the investigator
* Severe dyspnea at rest requiring supplementary oxygen therapy
* Severe uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 1999-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (36):
- Australia (6):
  - Liverpool, New South Wales
  - Waratah, New South Wales
  - Brisbane, Queensland
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Parkville, Victoria
- Brussels, Belgium
- Beijing, China
- Marseille, France
- Germany (7):
  - Berlin
  - Göttingen
  - Hamburg
  - Heidelberg
  - Lübeck
  - München
  - Trier
- Guatemala City, Guatemala
- Hungary (2):
  - Budapest
  - Debrecen
- Ramat Gan, Israel
- Auckland, New Zealand
- Panama City, Panama
- Gdansk, Poland
- Lisbon, Portugal
- Russia (3):
  - Izhevsk
  - Moscow
  - Saint Petersburg
- Belgrade, Serbia
- South Korea (2):
  - Bundang City
  - Seoul
- Spain (2):
  - Alicante, Alicante
  - Barcelona, Barcelona
- United Kingdom (4):
  - Edinburgh
  - Glasgow
  - London
  - Nottingham

REFERENCES:
- [Derived] Muller V, Clemens M, Jassem J, Al-Sakaff N, Auclair P, Nuesch E, Holloway D, Shing M, Bang YJ. Long-term trastuzumab (Herceptin(R)) treatment in a continuation study of patients with HER2-positive breast cancer or HER2-positive gastric cancer. BMC Cancer. 2018 Mar 15;18(1):295. doi: 10.1186/s12885-018-4183-2. PMID 29544445

RESULTS

PARTICIPANT FLOW:
Groups:
- Herceptin: Participants received intravenous (IV) Herceptin until disease progression, unacceptable toxicity, death, or decision by the investigator or participant to discontinue treatment. Herceptin was administered at the discretion of the investigator as either 2 milligrams per kilogram (mg/kg) once weekly (first dose as a 4-mg/kg loading dose) or 6 mg/kg every 3 weeks (first dose as an 8-mg/kg loading dose) via IV infusion over 90 minutes.
Period: Overall Study
Arm/Group | Herceptin
Started | 69
Completed | 69 (In this continued access study, all participants were considered to have completed per protocol.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Age was the only demographic variable collected for the study and was only collected from 32 participants. Gender, weight, and race were not collected under the protocol.
Groups:
- Herceptin: Participants received IV Herceptin until disease progression, unacceptable toxicity, death, or decision by the investigator or participant to discontinue treatment. Herceptin was administered at the discretion of the investigator as either 2 mg/kg once weekly (first dose as a 4-mg/kg loading dose) or 6 mg/kg every 3 weeks (first dose as an 8-mg/kg loading dose) via IV infusion over 90 minutes.
Arm/Group | Herceptin
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was the only demographic variable collected for the study and was only collected from 32 participants.
  years
    number analyzed (Participants) | 32
    (all) | 58.0 (11.00)
Sex/Gender, Customized [Number; unit: participants] — Population: Gender information was not collected under the protocol.

OUTCOME MEASURES:

1. Primary Outcome: On-Study Duration of Trial Treatment
Time Frame: From date of enrollment until death or premature withdrawal (maximum 7.4 years of follow-up)
Population: Analysis was performed on all enrolled participants.
Measure: Median (Full Range); unit: days
Arm/Group | Herceptin
Number analyzed (Participants) | 69
days | 386.0 [1 to 2697]

2. Primary Outcome: Number of Participants With Drop in Left Ventricular Ejection Fraction (LVEF) Below 45 Percent (%)
Time Frame: From date of enrollment until disease progression, death, or premature withdrawal; assessed per investigator discretion (maximum 7.4 years of follow-up)
Population: All enrolled participants with available LVEF data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Herceptin
Number analyzed (Participants) | 26
Participants | 0

3. Primary Outcome: Number of Participants Withdrawn From Study Because of LVEF Dysfunction
Description: LVEF dysfunction was defined as low LVEF measured on two consecutive assessments, with the second assessment performed after 3 weeks of study medication being withheld. Low LVEF included values less than or equal to 39% or values between 40% and 45% (inclusive) with a decrease of 10 or more percentage points from Baseline.
Time Frame: From date of enrollment until death or premature withdrawal (maximum 7.4 years of follow-up)
Population: All enrolled participants with available LVEF data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Herceptin
Number analyzed (Participants) | 26
Participants | 0

ADVERSE EVENTS:
Time Frame: From date of enrollment until disease progression, unacceptable toxicity, death, or decision by the investigator or participant to discontinue treatment (up to approximately 7.4 years)
Description: Only serious adverse events were collected during the trial. Terms were reported verbatim as provided by the reporter and were not re-coded. Analysis was performed on all enrolled participants.
Arm/Group | Herceptin
Serious Adverse Events (participants affected / at risk) | 11/69
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin (N=69)
Arthritis bacterial (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pain management (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.